CLINICAL TRIAL: NCT03243006
Title: Effect of Early Analgesic Treatment on Opioid Consumption
Brief Title: Effect of Early Pain Management at Triage on Opioid Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Triage treatment
Record Dates: First submitted 2017-07-15; First posted 2017-08-08 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Acute Pain
Keywords: acute pain; emergency department; opioid consumption
MeSH Terms: conditions — Acute Pain; Emergencies | interventions — Acetaminophen; Tramadol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group Placebo (Placebo Comparator): Patients in this group (Placebo Oral Tablet) received two placebo tablets
  Interventions: Drug: Placebo Oral Tablet
- group Paracetamol (Active Comparator): Patients in this group received two 500 mg paracetamol tablets
  Interventions: Drug: Paracetamol
- group Tramadol/Paracetamol combination (Active Comparator): Patients in this group (Tramadol/Paracetamol combination ) received 2 tablets of Tramadol/Paracetamol combination (37.5mg/325mg)
  Interventions: Drug: Tramadol/Paracetamol combination

INTERVENTIONS:
Drug: Paracetamol — 2 tablets of 500mg of paracetamol
  Arms: group Paracetamol
Drug: Tramadol/Paracetamol combination — 2 tablets of tramadol/paracetamol combination (32.5mg/325mg)
  Arms: group Tramadol/Paracetamol combination
Drug: Placebo Oral Tablet — 2 tablets of placebo
  Arms: group Placebo

SUMMARY:
introduction: Pain remains one of the most common reasons of emergency department admission. Opioids are overprescribed in emergency departments to treat severe pain.

objective: assessing the impact of ealy pain pain management on the use of intravenous morphine and on patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* a visual analog scale (VAS) equal to or higher than 30/100 ,
* having given consent to participation
* No contraindications to products used in the course of the study.

Exclusion Criteria:

* having a vital distress that does not allow an adequate assessment of the intensity of the pain
* an inability to assess pain intensity according to the VAS,
* swallowing disorders or inability , or a contraindication or an allergy to the treatments used.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
use of rescue opioids | DURING emergency department stay
  decreased consumption of intravenous morphine

SECONDARY OUTCOMES:
patient satisfaction | When quitting emergency department
  patient satisfaction regarding the overall management in the emergency department measured by likert scale
Length of emergency department stay | Until emergency department discharge
Pain intensity at emergency department discharge | At emergency department discharge
  Percentage of patients with visual analog scale <30

IPD SHARING:
Plan to Share IPD: Undecided